CLINICAL TRIAL: NCT00915343
Title: A, Randomised, Controlled, Two-armed, Two-period Cross-over, Multi-centre Phase II/III Study to Assess the Safety and Pharmacokinetics of Once-daily Oral Modified-release Hydrocortisone in Patients With Adrenal Insufficiency
Brief Title: Once-daily Oral Modified Release Hydrocortisone in Patients With Adrenal Insufficiency
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DC 06/02; 104-07; 2006-007084-89 (EudraCT Number)
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Adrenal Insufficiency
Keywords: Adrenal insufficiency; Primary adrenal insufficiency; Addison's disease; Hydrocortisone; Modified release
MeSH Terms: conditions — Adrenal Insufficiency; Addison Disease | interventions — Hydrocortisone; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Novel once daily modified release (Experimental): Test drug: hydrocortisone (modified release), oral tablet, available as 20 mg and 5 mg.
  The modified release hydrocortisone tablet was administered orally o.d. at 8 AM in the fasting state
  Interventions: Drug: hydrocortisone (modified release), oral tablet 20 and 5 mg
- Conventional TID hydrocortisone (Active Comparator): Reference drug: hydrocortisone, oral tablet, 10 mg. The reference drug was administered orally thrice daily (at 8 AM, 12 AM and 4 PM)in the same total daily dose as the experimental drug. The morning dose was administered in the fasting state.
  Interventions: Drug: Hydrocortisone, oral tablet, 10 mg

INTERVENTIONS:
Drug: hydrocortisone (modified release), oral tablet 20 and 5 mg — The modified release hydrocortisone tablet was administered orally o.d. at 8 AM in the fasting state. The dose was the same as patients have had before entering the trial
  Other Names: DuoCort
  Arms: Novel once daily modified release
Drug: Hydrocortisone, oral tablet, 10 mg — The reference drug was administered orally thrice daily (at 8 AM, 12 AM and 4 PM). The morning dose was administered in the fasting state. The total daily dose was the same as in the experimental treatment arm.
  Arms: Conventional TID hydrocortisone

SUMMARY:
This is a randomised, controlled, open, two-armed, two-period cross-over, multi-centre phase II/III study to assess the safety, tolerability and pharmacokinetics of once-daily oral modified-release hydrocortisone in comparison to conventional thrice-daily oral hydrocortisone tablets in patients with adrenal insufficiency

DETAILED DESCRIPTION:
Adrenal insufficiency is a disease with more than 80% 1-year mortality before the availability of synthetic glucocorticoids. Current replacement therapy has improved this dramatically, but recent data suggest that outcome is still compromised. Patient receiving replacement therapy with hydrocortisone or cortisone acetate have compromised quality of life, reduced bone mass, increased risk factors for cardiovascular disease and premature mortality that is more than twice the mortality rate in the background population.

Circulating cortisol levels follow a distinct diurnal pattern with high levels in the early morning and low trough values around midnight. Using available formulations for replacement therapy this circadian rhythm is had to mimic and also during the active time of the day high peaks and low troughs occur.

In this trial a newly developed novel dual-, controlled release formulation of hydrocortisone that has in healthy volunteers been able to mimic the circadian pattern of circulating cortisol was studied in patients with primary adrenal insufficiency (Addison's disease).

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed (e.g. more than 6 months ago) primary adrenal insufficiency with a stable daily glucocorticoid substitution dose for at least 3 months prior to study entry
* Signed informed consent to participate in the study.

Exclusion Criteria:

* Clinical or laboratory signs of significant cerebral, cardiovascular, respiratory, Hepatobiliary, pancreatic disease
* Clinically significant renal dysfunction
* Clinical or laboratory signs of significant gastrointestinal emptying or motility disease
* Any medication with agents which could interfere with hydrocortisone kinetics
* Pregnant or lactating women
* Regular dehydroepiandrosterone (DHEA) medication for the past 4 weeks
* Oral oestrogen medication for the past 4 weeks
* Deranged mineralocorticoid status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-08-21 (Actual); Primary Completion 2008-07-28 (Actual); Study Completion 2009-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Forss, MSc BA, Study Director — DuoCort AB; Anna G Nilsson, MD, PhD, Principal Investigator — Göteborg University

REFERENCES:
- [Background] Johannsson G, Bergthorsdottir R, Nilsson AG, Lennernas H, Hedner T, Skrtic S. Improving glucocorticoid replacement therapy using a novel modified-release hydrocortisone tablet: a pharmacokinetic study. Eur J Endocrinol. 2009 Jul;161(1):119-30. doi: 10.1530/EJE-09-0170. Epub 2009 Apr 21. PMID 19383806
- [Background] Lennernas H, Skrtic S, Johannsson G. Replacement therapy of oral hydrocortisone in adrenal insufficiency: the influence of gastrointestinal factors. Expert Opin Drug Metab Toxicol. 2008 Jun;4(6):749-58. doi: 10.1517/17425255.4.6.749. PMID 18611115
- [Background] Esteban NV, Loughlin T, Yergey AL, Zawadzki JK, Booth JD, Winterer JC, Loriaux DL. Daily cortisol production rate in man determined by stable isotope dilution/mass spectrometry. J Clin Endocrinol Metab. 1991 Jan;72(1):39-45. doi: 10.1210/jcem-72-1-39. PMID 1986026
- [Background] Filipsson H, Monson JP, Koltowska-Haggstrom M, Mattsson A, Johannsson G. The impact of glucocorticoid replacement regimens on metabolic outcome and comorbidity in hypopituitary patients. J Clin Endocrinol Metab. 2006 Oct;91(10):3954-61. doi: 10.1210/jc.2006-0524. Epub 2006 Aug 8. PMID 16895963
- [Background] Suliman AM, Freaney R, Smith TP, McBrinn Y, Murray B, McKenna TJ. The impact of different glucocorticoid replacement schedules on bone turnover and insulin sensitivity in patients with adrenal insufficiency. Clin Endocrinol (Oxf). 2003 Sep;59(3):380-7. doi: 10.1046/j.1365-2265.2003.01860.x. PMID 12919163
- [Background] Feek CM, Ratcliffe JG, Seth J, Gray CE, Toft AD, Irvine WJ. Patterns of plasma cortisol and ACTH concentrations in patients with Addison's disease treated with conventional corticosteroid replacement. Clin Endocrinol (Oxf). 1981 May;14(5):451-8. doi: 10.1111/j.1365-2265.1981.tb00634.x. PMID 6273020
- [Background] Howlett TA. An assessment of optimal hydrocortisone replacement therapy. Clin Endocrinol (Oxf). 1997 Mar;46(3):263-8. doi: 10.1046/j.1365-2265.1997.1340955.x. PMID 9156032
- [Background] Groves RW, Toms GC, Houghton BJ, Monson JP. Corticosteroid replacement therapy: twice or thrice daily? J R Soc Med. 1988 Sep;81(9):514-6. doi: 10.1177/014107688808100906. PMID 3184107
- [Background] Lovas K, Gjesdal CG, Christensen M, Wolff AB, Almas B, Svartberg J, Fougner KJ, Syversen U, Bollerslev J, Falch JA, Hunt PJ, Chatterjee VK, Husebye ES. Glucocorticoid replacement therapy and pharmacogenetics in Addison's disease: effects on bone. Eur J Endocrinol. 2009 Jun;160(6):993-1002. doi: 10.1530/EJE-08-0880. Epub 2009 Mar 12. PMID 19282465
- [Background] al-Shoumer KA, Beshyah SA, Niththyananthan R, Johnston DG. Effect of glucocorticoid replacement therapy on glucose tolerance and intermediary metabolites in hypopituitary adults. Clin Endocrinol (Oxf). 1995 Jan;42(1):85-90. doi: 10.1111/j.1365-2265.1995.tb02602.x. PMID 7889636
- [Background] Hahner S, Loeffler M, Fassnacht M, Weismann D, Koschker AC, Quinkler M, Decker O, Arlt W, Allolio B. Impaired subjective health status in 256 patients with adrenal insufficiency on standard therapy based on cross-sectional analysis. J Clin Endocrinol Metab. 2007 Oct;92(10):3912-22. doi: 10.1210/jc.2007-0685. Epub 2007 Aug 7. PMID 17684047
- [Background] Bergthorsdottir R, Leonsson-Zachrisson M, Oden A, Johannsson G. Premature mortality in patients with Addison's disease: a population-based study. J Clin Endocrinol Metab. 2006 Dec;91(12):4849-53. doi: 10.1210/jc.2006-0076. Epub 2006 Sep 12. PMID 16968806
- [Background] Dallman MF, Akana SF, Bhatnagar S, Bell ME, Strack AM. Bottomed out: metabolic significance of the circadian trough in glucocorticoid concentrations. Int J Obes Relat Metab Disord. 2000 Jun;24 Suppl 2:S40-6. doi: 10.1038/sj.ijo.0801276. PMID 10997607
- [Derived] Espiard S, McQueen J, Sherlock M, Ragnarsson O, Bergthorsdottir R, Burman P, Dahlqvist P, Ekman B, Engstrom BE, Skrtic S, Wahlberg J, Stewart PM, Johannsson G. Improved Urinary Cortisol Metabolome in Addison Disease: A Prospective Trial of Dual-Release Hydrocortisone. J Clin Endocrinol Metab. 2021 Mar 8;106(3):814-825. doi: 10.1210/clinem/dgaa862. PMID 33236103

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study consisted of Part A (cross-over) and Part B (open-label). Of the 64 participants started and completed Part A, 5 participants did not enter Part B (treatment switch=2, withdrawal by participant= 2, nausea and abnormal laboratory value=1), 59 started Part B of the study.
Groups:
- Hydrocortisone MR OD Then Hydrocortisone TID - Part A: Participants received novel once daily (OD) hydrocortisone modified release (MR) tablets in the first intervention period then hydrocortisone tablets thrice daily (TID) in the second intervention period, at the same total daily dose of 20 to 40 milligram (mg) for 12 weeks.
- Hydrocortisone TID Then Hydrocortisone MR OD - Part A: Participants received hydrocortisone tablets TID in the first intervention period then novel OD hydrocortisone MR tablets in the second intervention period, at the same total daily dose of 20 to 40 mg for 12 weeks.
- Hydrocortisone MR Tablet OD - Part B (All 6 Months): Hydrocortisone MR tablets 20 to 40 mg orally OD for 6 months.
Period: Part A - First Intervention Period
Arm/Group | Hydrocortisone MR OD Then Hydrocortisone TID - Part A | Hydrocortisone TID Then Hydrocortisone MR OD - Part A | Hydrocortisone MR Tablet OD - Part B (All 6 Months)
Started | 32 | 32 | 0
Completed | 32 | 32 | 0
Not Completed | 0 | 0 | 0
Period: Part A - Second Intervention Period
Arm/Group | Hydrocortisone MR OD Then Hydrocortisone TID - Part A | Hydrocortisone TID Then Hydrocortisone MR OD - Part A | Hydrocortisone MR Tablet OD - Part B (All 6 Months)
Started | 32 | 32 | 0
Completed | 32 | 32 | 0
Not Completed | 0 | 0 | 0
Period: Part B - Open Label Period
Arm/Group | Hydrocortisone MR OD Then Hydrocortisone TID - Part A | Hydrocortisone TID Then Hydrocortisone MR OD - Part A | Hydrocortisone MR Tablet OD - Part B (All 6 Months)
Started | 0 | 0 | 59
Completed | 0 | 0 | 57
Not Completed | 0 | 0 | 2
Not completed — Treatment switch | 0 | 0 | 1
Not completed — Did not attend the last visit | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention-To-Treat (ITT) set included all randomised participants who took at least 1 dose of study drug with assessments of any variables or with primary efficacy assessments including all pharmacokinetic (PK) samplings during any of the treatment periods.
Groups:
- Entire Study: Included all participants randomized to receive hydrocortisone MR tablets orally OD first or hydrocortisone tablets orally TID first; in any of the intervention periods during the 12-week cross-over period of Part A or hydrocortisone MR tablets orally OD during the 6-month open-label period of Part B.
Arm/Group | Entire Study
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 37

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Time Curve From Zero to 24 Hours (AUC0-24h) of Total S-cortisol in Plasma After Multiple Doses During Part A
Description: AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body. Participants in Arm 1 underwent standardised in-house PK sampling during 24 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The data for combined arm 1+2 after multiple doses were reported.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A: Intention-To-Treat (ITT) set included all randomised participants who took at least 1 dose of study drug with primary efficacy assessments including all pharmacokinetic (PK) samplings during either treatment period. Here "number of participants analysed" signifies those who were evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: hour*nanomole per liter
Groups:
- Hydrocortisone MR Tablet OD - Part A: Hydrocortisone MR tablets 20 to 40 mg orally OD during Part A of the study.
- Hydrocortisone Tablet TID - Part A: Hydrocortisone tablets 20 to 40 mg orally TID during Part A of the study.
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 59 | 59
hour*nanomole per liter | 3962.0 (1079.6) | 4879.6 (1194.4)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p < 0.0001, ANOVA — Comparison of log S-cortisol AUC between OD and TID regimens was adjusted for both period effect and subject effect using generalized linear model (GLM) in statistical analysis system (SAS); Period-adjusted quotient = 0.806, 95% CI 2-sided [0.753 to 0.862] — The quotient was defined as AUC0-24h for OD treatment divided by AUC0-24h for TID treatment

2. Secondary Outcome: Maximal Concentration (Cmax1) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated. Cmax1 is the Cmax after first dose of study drug. Participants in Arm 1 underwent standardised in-house PK sampling during 24 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The average of single and multiple dosing for combined arm 1+2 was reported.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: nanomoles per liter
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 61 | 61
nanomoles per liter | 690.7 (109.2) | 802.8 (136.2)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test; Mean difference = -111.989, 95% CI 2-sided [-133.980 to 89.999]

3. Secondary Outcome: Maximal Concentration (Cmax2) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated. Cmax2 is the Cmax after second dose of study drug. Participants in Arm 1 underwent standardised in-house PK sampling during 24 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The average of single and multiple dosing for combined arm 1+2 was reported.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: nanomoles per liter
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 8 | 8
nanomoles per liter | 553.8 (170.8) | 446.9 (129.3)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p = 0.0357, Fisher's non-parametric permutation test; Mean difference = 110.417, 95% CI 2-sided [16.755 to 204.078]

4. Secondary Outcome: Average Concentration of S-cortisol During the Dosing Interval at Steady State (Css,av) in Plasma After Single and Multiple Dosing During Part A
Description: Css,av was calculated as the area under the S-cortisol concentration versus time curve during a dosing interval at steady state (AUCtau) divided by dosing interval (tau). Participants in Arm 1 underwent standardised in-house PK sampling during 24 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The average of single and multiple dosing for combined arm 1+2 was reported.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: nanomoles per liter
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 59 | 59
nanomoles per liter | 165.1 (45.0) | 203.3 (49.8)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test; Mean difference = -38.076, 95% CI 2-sided [-50.276 to 25.876]

5. Secondary Outcome: First Detectable Concentration (Cfirst) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: Participants in Arm 1 underwent standardised in-house PK sampling during 24 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The average of single and multiple dosing for combined arm 1+2 was reported.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: nanomoles per liter
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 62 | 62
nanomoles per liter | 229.0 (169.8) | 295.1 (203.2)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p = 0.0033, Fisher's non-parametric permutation test; Mean difference = -65.782, 95% CI 2-sided [-109.201 to 22.362]

6. Secondary Outcome: Concentration at 6 Hours (C6h) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: as for outcome 5
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: nanomoles per liter
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 60 | 60
nanomoles per liter | 278.5 (134.9) | 426.7 (135.2)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test; Mean difference = -148.015, 95% CI 2-sided [-189.469 to -106.561]

7. Secondary Outcome: Concentration at 7 Hours (C7h) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: as for outcome 5
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: nanomoles per liter
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 60 | 60
nanomoles per liter | 214.1 (106.8) | 322.4 (110.0)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test; Mean difference = -108.306, 95% CI 2-sided [-140.193 to -76.420]

8. Secondary Outcome: Time to Peak Plasma Concentration (Tmax1) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: Tmax is the time after administration of a drug when the maximum plasma concentration in the body is reached. Tmax1 is the Tmax after first dose of study drug. Participants in Arm 1 underwent standardised in-house PK sampling during 24 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The average of single and multiple dosing for combined arm 1+2 was reported.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 61 | 61
hours | 1.00 [0.38 to 5.00] | 0.750 [0.292 to 2.750]
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p = 0.0214, Fisher's non-parametric permutation test; Mean difference = 0.270, 95% CI 2-sided [0.028 to 0.512]

9. Secondary Outcome: Time to Peak Plasma Concentration (Tmax2) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: Tmax is the time after administration of a drug when the maximum plasma concentration in the body is reached. Tmax2 is the Tmax after second dose of study drug. Participants in Arm 1 underwent standardised in-house PK sampling during 24 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The average of single and multiple dosing for combined arm 1+2 was reported.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 8 | 8
hours | 5.00 [3.50 to 6.00] | 6.00 [5.00 to 6.00]
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p = 0.0714, Fisher's non-parametric permutation test; Mean difference = -1.042, 95% CI 2-sided [-2.098 to 0.015]

10. Secondary Outcome: Time to First Detectable Concentration (Tfirst) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: as for outcome 5
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 62 | 62
hours | 0.229 [0.000 to 0.625] | 0.208 [0.000 to 0.500]
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p = 0.6687, Fisher's non-parametric permutation test; Mean difference = -0.007, 95% CI 2-sided [-0.038 to 0.024]

11. Secondary Outcome: Time to Reach a Concentration of 200 Nanometers (nM) (T200) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: as for outcome 5
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 62 | 62
hours | 0.250 [0.000 to 0.750] | 0.167 [0.063 to 0.563]
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p = 0.0280, Fisher's non-parametric permutation test; Mean difference = 0.049, 95% CI 2-sided [0.006 to 0.093]

12. Secondary Outcome: Drug Concentration Half-Life From 5 to 24 Hours (t1/2[5-24h]) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: t1/2[5-24h] is the time taken for the blood plasma concentration of a drug to halve from 5 to 24 hours. Participants in Arm 1 underwent standardised in-house PK sampling during 24 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The average of single and multiple dosing for combined arm 1+2 was reported.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 17 | 17
hours | 7.32 (9.32) | 1.84 (0.93)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p = 0.0003, Fisher's non-parametric permutation test; Mean difference = 5.509, 95% CI 2-sided [0.751 to 10.268]

13. Secondary Outcome: Drug Concentration Half-Life From 5 to 14 Hours (t1/2[5-14h]) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: t1/2[5-14h] is the time taken for the blood plasma concentration of a drug to halve from 5 to 14 hours. Participants in Arm 1 underwent standardised in-house PK sampling during 24 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The average of single and multiple dosing for combined arm 1+2 was reported.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 52 | 52
hours | 4.60 (5.82) | 18.4 (24.5)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test; Mean difference = -13.800, 95% CI 2-sided [-20.533 to -7.067]

14. Secondary Outcome: Area Under the Concentration Time Curve (AUC) Between Specified Timepoints of Total S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body. AUC between specified timepoints included AUC0-4h, AUC4-12h, AUC6-12h, AUC12-24h, AUC0-10h, AUC4-10h, AUC6-10h, AUC10-24h, AUC(0-inf), AUC(24h-inf). Participants in Arm 1 underwent standardised in-house PK sampling during 24 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The average of single and multiple dosing for combined arm 1+2 was reported. Here, "N"signifies the number of participants evaluable for this outcome.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population.
Measure: Mean (Standard Deviation); unit: hour*nanomole per liter
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 63 | 63
hour*nanomole per liter
  AUC0-4h (N=61, 61) | 2053.7 (432.0) | 1929.7 (409.9)
  AUC4-12h (N=61, 61) | 1491.8 (638.9) | 2302.5 (669.3)
  AUC6-12h (N=61, 61) | 808.2 (386.3) | 1607.6 (483.3)
  AUC12-24h (N=61, 61) | 306.2 (305.2) | 576.6 (681.6)
  AUC0-10h (N=61, 61) | 3388.4 (915.0) | 3768.7 (968.5)
  AUC4-10h (N=61, 61) | 1334.7 (582.5) | 1839.0 (599.0)
  AUC6-10h (N=61, 61) | 651.1 (322.1) | 1144.1 (404.6)
  AUC10-24h (N=61, 61) | 465.0 (352.2) | 1058.0 (752.4)
  AUC(0-inf) (N=52, 52) | 3972.6 (1125.9) | 5162.8 (1777.2)
  AUC(24h-inf) (N=52, 52) | 195.3 (568.1) | 410.4 (1094.0)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; AUC0-4h; Test type: Superiority or Other; p = 0.0002, ANOVA; Period-adjusted quotient = 1.064, 95% CI 2-sided [1.032 to 1.097] — The quotient was defined as AUC0-4h for OD treatment divided by AUC0-4h for TID treatment
Statistical Analysis 2: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; AUC4-12h; Test type: Superiority or Other; p < 0.0001, ANOVA; Period-adjusted quotient = 0.617, 95% CI 2-sided [0.563 to 0.675] — The quotient was defined as AUC4-12h for OD treatment divided by AUC4-12h for TID treatment
Statistical Analysis 3: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; AUC6-12h; Test type: Superiority or Other; p < 0.0001, ANOVA; Period-adjusted quotient = 0.472, 95% CI 2-sided [0.424 to 0.525] — The quotient was defined as AUC6-12h for OD treatment divided by AUC6-12h for TID treatment
Statistical Analysis 4: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; AUC12-24h; Test type: Superiority or Other; p = 0.0003, ANOVA; Period-adjusted quotient = 0.588, 95% CI 2-sided [0.446 to 0.775] — The quotient was defined as AUC12-24h for OD treatment divided by AUC12-24h for TID treatment
Statistical Analysis 5: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; AUC0-10h; Test type: Superiority or Other; p < 0.0001, ANOVA; Period-adjusted quotient = 0.894, 95% CI 2-sided [0.856 to 0.935] — The quotient was defined as AUC0-10h for OD treatment divided by AUC0-10h for TID treatment
Statistical Analysis 6: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; AUC4-10h; Test type: Superiority or Other; p < 0.0001, ANOVA; Period-adjusted quotient = 0.695, 95% CI 2-sided [0.632 to 0.765] — The quotient was defined as AUC4-10h for OD treatment divided by AUC4-10h for TID treatment
Statistical Analysis 7: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; AUC6-10h; Test type: Superiority or Other; p < 0.0001, ANOVA; Period-adjusted quotient = 0.540, 95% CI 2-sided [0.482 to 0.605] — The quotient was defined as AUC6-10h for OD treatment divided by AUC6-10h for TID treatment
Statistical Analysis 8: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; AUC10-24h; Test type: Superiority or Other; p < 0.0001, ANOVA; Period-adjusted quotient = 0.412, 95% CI 2-sided [0.338 to 0.504] — The quotient was defined as AUC10-24h for OD treatment divided by AUC10-24h for TID treatment
Statistical Analysis 9: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; AUC(0-inf); Test type: Superiority or Other; p < 0.0001, ANOVA; Period-adjusted quotient = 0.776, 95% CI 2-sided [0.714 to 0.843] — The quotient was defined as AUC(0-inf) for OD treatment divided by AUC(0-inf) for TID treatment
Statistical Analysis 10: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; AUC(24h-inf); Test type: Superiority or Other; p = 0.8770, ANOVA; Period-adjusted quotient = 1.069, 95% CI 2-sided [0.453 to 2.521] — The quotient was defined as AUC(24h-inf) for OD treatment divided by AUC(24h-inf) for TID treatment

15. Secondary Outcome: Area Under the Concentration Time Curve During a Dosing Interval at Steady State (AUCtau) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body. AUCtau is defined as AUC during a dosing interval at steady state. Participants in Arm 1 underwent standardised in-house PK sampling during 24 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The average of single and multiple dosing for combined arm 1+2 was reported.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: hour*nanomole per liter
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 59 | 59
hour*nanomole per liter | 3962.0 (1079.6) | 4879.6 (1194.4)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p < 0.0001, ANOVA; Period-adjusted quotient = 0.806, 95% CI 2-sided [0.753 to 0.862] — The quotient was defined as AUCtau for OD treatment divided by AUCtau for TID treatment

16. Secondary Outcome: Area Under the Concentration Time Curve During a Dosing Interval at Steady State Adjusted by Dose (AUCtau/Dose) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body. Participants in Arm 1 underwent standardised in-house PK sampling during 14 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The average of single and multiple dosing for combined arm 1+2 was reported.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: hour per liter
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 59 | 59
hour per liter | 0.048 (0.016) | 0.061 (0.017)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p < 0.0001, ANOVA; Period-adjusted quotient = 0.790, 95% CI 2-sided [0.734 to 0.851] — The quotient was defined as AUCtau/dose for OD treatment divided by AUCtau/dose for TID treatment

17. Secondary Outcome: Area Under the Concentration Time Curve From Zero to 24 Hours Adjusted by Dose (AUC0-24h/Dose) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body. Participants in Arm 1 underwent standardised in-house PK sampling during 24 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The average of single and multiple dosing for combined arm 1+2 was reported.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: hour per liter
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 61 | 61
hour per liter | 0.047 (0.014) | 0.060 (0.018)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p < 0.0001, ANOVA; Period-adjusted quotient = 0.785, 95% CI 2-sided [0.741 to 0.831] — The quotient was defined as AUC0-24h/dose for OD treatment divided by AUC0-24h/dose for TID treatment

18. Secondary Outcome: Area Under the Concentration Time Curve From Zero to 10 Hours Adjusted by Dose (AUC0-10h/Dose) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: as for outcome 17
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: hour per liter
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 61 | 61
hour per liter | 0.041 (0.012) | 0.046 (0.013)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p < 0.0001, ANOVA; Period-adjusted quotient = 0.885, 95% CI 2-sided [0.844 to 0.926] — The quotient was defined as AUC0-10h/dose for OD treatment divided by AUC0-10h/dose for TID treatment

19. Secondary Outcome: Area Under the Concentration Time Curve From Zero to 4 Hours Adjusted by Dose (AUC0-4h/Dose) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: as for outcome 17
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: hour per liter
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 61 | 61
hour per liter | 0.025 (0.005) | 0.024 (0.006)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p = 0.0020, ANOVA; Period-adjusted quotient = 1.053, 95% CI 2-sided [1.020 to 1.086] — The quotient was defined as AUC0-4h/dose for OD treatment divided by AUC0-4h/dose for TID treatment

20. Secondary Outcome: Average Concentration of S-cortisol During the Dosing Interval at Steady State Adjusted by Dose (Css,av/Dose) in Plasma After Single and Multiple Dosing During Part A
Description: as for outcome 4
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: per liter
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 59 | 59
per liter | 0.002 (0.001) | 0.003 (0.001)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test; Mean difference = -0.001, 95% CI 2-sided [-0.001 to -0.000]

21. Secondary Outcome: Maximal Concentration Adjusted by Dose (Cmax1/Dose) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: as for outcome 2
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: per liter
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 61 | 61
per liter | 0.008 (0.002) | 0.010 (0.002)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p < 0.0001, Fisher's non-parametric permutation test; Mean difference = -0.001, 95% CI 2-sided [-0.002 to -0.001]

22. Secondary Outcome: Time to First Detectable Concentration Adjusted by Dose (Tfirst/Dose) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: as for outcome 5
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: (hour per nanomole)*10^6
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 62 | 62
(hour per nanomole)*10^6 | 2.26 (1.69) | 2.32 (1.43)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p = 0.7827, Fisher's non-parametric permutation test; Mean difference = -0.055, 95% CI 2-sided [-0.444 to 0.334]

23. Secondary Outcome: First Detectable Concentration Adjusted by Dose (Cfirst/Dose) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: as for outcome 5
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: per liter
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 62 | 62
per liter | 0.003 (0.002) | 0.004 (0.002)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p = 0.0015, Fisher's non-parametric permutation test; Mean difference = -0.001, 95% CI 2-sided [-0.001 to -0.000]

24. Secondary Outcome: Percentage (%) of Area Under the Concentration Time Curve (AUC) Extrapolation of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: The percentage of AUC0-inf that is due to extrapolation from Tlast to infinity (AUC%Extrapolation) was calculated by using the formula AUC%extrapolation = 100*(AUC0-inf minus AUC0-t)/AUC0-inf. The function of this parameter was to provide information about what percentage of the theoretical curve (AUC0-inf) was possible to determine experimentally (AUC0-t). Therefore, on average, it is expected that the residual area (AUCextrapolation) is not greater than 20%. Participants in Arm 1 underwent standardised in-house PK sampling during 24 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The average of single and multiple dosing for combined arm 1+2 was reported.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: percentage of AUC
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 52 | 52
percentage of AUC | 10.1 (7.9) | 9.26 (12.74)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p < 0.0001, ANOVA; Period-adjusted quotient = 6.098, 95% CI 2-sided [2.940 to 12.646] — The quotient was defined as AUC Extrapolation for OD treatment divided by AUC Extrapolation for TID treatment

25. Secondary Outcome: Percentage (%) of Fluctuation in Concentrations of S-cortisol at Steady State in Plasma After Single and Multiple Dosing During Part A
Description: Percentage of fluctuation was calculated by using formula 100*(Cmax-minimum plasma concentration [Cmin])/Cavg,ss. It was peak trough fluctuation within one dosing interval at steady state. Participants in Arm 1 underwent standardised in-house PK sampling during 24 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The average of single and multiple dosing for combined arm 1+2 was reported.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: percentage of fluctuation
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 59 | 59
percentage of fluctuation | 429.7 (117.3) | 396.2 (99.0)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p = 0.0396, Fisher's non-parametric permutation test; Mean difference = 33.532, 95% CI 2-sided [1.734 to 65.329]

26. Secondary Outcome: Accumulation Ratio (Rac) of S-cortisol in Plasma After Single and Multiple Dosing During Part A
Description: The Rac was calculated as area under the S-cortisol concentration versus time curve during a dosing interval at steady state (AUCtau) on Day 28 divided by AUC0-24h on Day 1. Participants in Arm 1 underwent standardised in-house PK sampling during 24 hours in order to assess single-dose PK of OD or TID regimen at the start of each study treatment period while participants in Arm 2 had a reduced PK sampling scheme of single dose PK on Days 1-2 and returned for multiple-dose PK sampling on Days 7-8. The average of single and multiple dosing for combined arm 1+2 was reported.
Time Frame: Arm 1: Week 4, Week 16, Week 16 + 1 day, Week 28; Arm 2: Week 4, Week 4 + 7 days, Week 16, Week 16 + 7 days
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 55 | 55
ratio | 1.11 (0.29) | 1.03 (0.19)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p = 0.1032, Fisher's non-parametric permutation test; Period-adjusted quotient = 0.080, 95% CI 2-sided [-0.017 to 0.177]

27. Secondary Outcome: Comparison of Overall Patient Tolerability Score Between Once Daily and Thrice Daily Therapy, Assessed by Patient and Investigator - Part A
Description: Overall patient tolerability score assessed by patient and investigator, ranged from 1 (feeling poor on treatment) to 5 (feeling very well on treatment). The average total score ranges from 1 to 5 with a higher score representing better tolerability of the treatment. Questionnaire assessed by patient were "I have been very poorly on the treatment", "I haven't been very well (or less well) on the treatment", "I have been acceptably well on the treatment", "I have been well on the treatment" and "I have been very well on the treatment". Questionnaire assessed by investigator were "The patient has been feeling very poorly on the treatment", "The patient has not tolerated the treatment well", "The patient has tolerated the treatment less well", "The patient has tolerated the treatment well" and "The patient has tolerated the treatment very well".
Time Frame: 12 weeks
Population: Part A ITT population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 63 | 63
scores on a scale
  Patient | 4.28 (0.74) | 4.36 (0.73)
  Investigator | 4.26 (0.73) | 4.33 (0.73)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Patient; Test type: Superiority or Other; p = 0.3767, Fisher's test; Fisher's non; least square mean = -0.078, 95% CI 2-sided [-0.250 to 0.094]
Statistical Analysis 2: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Investigator; Test type: Superiority or Other; p = 0.4625, Fisher's test; Fisher's non; least square mean = -0.064, 95% CI 2-sided [-0.235 to 0.107]

28. Secondary Outcome: Percentage (%) of Participants With Change From Baseline in Patient Tolerability Questionnaire at Month 6, Assessed by Patient and Investigator - Part B
Description: Patient tolerability questionnaire was assessed by both patient and investigator, the responses were as follows: improvement, no change, worsening and were reported.
Time Frame: Baseline (week 0), month 6
Population: Part B ITT population with participants evaluable for this outcome.
Measure: Number; unit: percentage of participants
Groups:
- Hydrocortisone MR Tablet OD - Part B (All 6 Months): Hydrocortisone MR tablets 20 to 40 mg orally OD during the entire 6-month period of Part B.
Arm/Group | Hydrocortisone MR Tablet OD - Part B (All 6 Months)
Number analyzed (Participants) | 56
percentage of participants
  Improvement (Patient) | 10.7
  Improvement (Investigator) | 14.0
  No change (Patient) | 73.2
  No change (Investigator) | 70.0
  Worsening (Patient) | 16.1
  Worsening (Investigator) | 16.0
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part B (All 6 Months); Patient; Test type: Superiority or Other; p = 0.6072, Sign test
Statistical Analysis 2: Comparison: Hydrocortisone MR Tablet OD - Part B (All 6 Months); Investigator; Test type: Superiority or Other; p = 1.0000, Sign test

29. Secondary Outcome: Comparison of Quality of Life (QoL) Assessed by Short Form-36 Survey (SF-36) For Physical and Mental Component Score Between Once Daily and Thrice Daily Therapy- Part A
Description: The SF-36 was a questionnaire used to assess physical functioning and is made up of eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health. Transforming and standardizing these domains lead to the calculation of the physical and mental component summary measures. Scores ranging from 0 to 100, with 0=worst score (or quality of life) and 100=best score. A higher value corresponds to better well-being.
Time Frame: 12 weeks
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 61 | 61
scores on a scale
  Physical component | 49.3 (9.1) | 50.0 (9.9)
  Mental component | 51.1 (7.3) | 49.8 (9.3)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Comparison of Quality of Life (QoL) Assessed by Short Form-36 Survey (SF-36) For Physical Component Score; Test type: Superiority or Other; p = 0.3332, Fisher's test; Fisher's non-parametric two-sample permutation test; Mean difference = -0.6
Statistical Analysis 2: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Comparison of Quality of Life (QoL) Assessed by Short Form-36 Survey (SF-36) For Mental Component Score; Test type: Superiority or Other; p = 0.3405, Fisher's test; Fisher's non-parametric two-sample permutation test; Mean difference = 0.9

30. Secondary Outcome: Change From Baseline to 6 Months in Quality of Life (QoL) Assessed by Short Form-36 Survey (SF-36) For Physical and Mental Component Score - Part B
Description: The SF-36 was a questionnaire used to assess physical functioning and is made up of eight domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health. Transforming and standardizing these domains lead to the calculation of the physical and mental component summary measures. Scores ranging from 0 to 100, with 0=worst score (or quality of life) and 100=best score. A higher value in the SF-36 questionnaire corresponds to better well-being.
Time Frame: Baseline (week 0), month 6
Population: Part B ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Hydrocortisone MR Tablet OD - Part B (All 6 Months)
Number analyzed (Participants) | 54
scores on a scale
  Physical component | 0.390 (4.374)
  Mental component | -0.896 (5.913)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part B (All 6 Months); Change From Baseline to 6 months in Quality of Life (QoL) Assessed by Short Form-36 Survey (SF-36) For Physical Component Score; Test type: Superiority or Other; p = 0.8418, Wilcoxon Signed Rank
Statistical Analysis 2: Comparison: Hydrocortisone MR Tablet OD - Part B (All 6 Months); Change From Baseline to 6 months in Quality of Life (QoL) Assessed by Short Form-36 Survey (SF-36) For Mental Component Score; Test type: Superiority or Other; p = 0.3550, Wilcoxon Signed Rank test

31. Secondary Outcome: Comparison of Quality of Life (QoL) Assessed by Fatigue Impact Scale (FIS) Total Score Between Once Daily and Thrice Daily Therapy - Part A
Description: FIS is a subject-reported scale that qualifies the impact of fatigue on daily life in participants. It consisted of 40 statements that measure fatigue in 3 areas: physical, cognitive, and psychosocial. This 40-item scale evaluates the construct of perceived impact of fatigue on everyday life. Respondents rated each statement using a 5-point Likert-type scale ranging from 0 (no problem) to 4 (extreme problem). A total score ranged from 0 to 160. A lower value corresponds to better well-being.
Time Frame: 12 weeks
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 62 | 61
scores on a scale | 22.6 (25.4) | 26.4 (30.3)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p = 0.0823, Fisher's; Fisher's non-parametric two-sample permutation test; Mean difference = -2.9

32. Secondary Outcome: Change From Baseline to 6 Months in Quality of Life (QoL) Assessed by Fatigue Impact Scale (FIS) Total Score - Part B
Description: as for outcome 31
Time Frame: Baseline (week 0), month 6
Population: Part B ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Hydrocortisone MR Tablet OD - Part B (All 6 Months)
Number analyzed (Participants) | 56
scores on a scale | -1.09 (12.49)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part B (All 6 Months); Test type: Superiority or Other; p = 0.5982, Wilcoxon Signed Rank test

33. Secondary Outcome: Comparison of Quality of Life (QoL) Assessed by Psychological General Well Being (PGWB) Total Scores Between Once Daily and Thrice Daily Therapy- Part A
Description: The PGWB consists of 22 self-administered items rated on a scale from 1 (worst level of well-being) to 6 (maximum level of well-being) with a total score ranging from 22 to 132. A higher score represents better well-being.
Time Frame: 12 weeks
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 62 | 61
scores on a scale | 110.5 (14.0) | 107.7 (17.3)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p = 0.0632, Fisher's test; Fisher's non-parametric two-sample permutation test; Mean difference = 2.3

34. Secondary Outcome: Change From Baseline to 6 Months in Quality of Life (QoL) Assessed by Psychological General Well Being (PGWB) Total Scores- Part B
Description: as for outcome 33
Time Frame: Baseline (week 0), month 6
Population: Part B ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Hydrocortisone MR Tablet OD - Part B (All 6 Months)
Number analyzed (Participants) | 55
scores on a scale | -0.739 (9.687)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part B (All 6 Months); Test type: Superiority or Other; p = 0.8676, Wilcoxon Signed Rank test

35. Secondary Outcome: Change From Baseline to 12 Weeks in Diurnal Fatigue Questionnaire for Day Average of Once Daily Therapy - Part A
Description: Diurnal fatigue was assessed at 8 ante meridian (AM), at 12 AM and at 4 post meridian (PM) by a visual analogue scale (VAS) based on 8 domains (energy, relaxed, less alert, moody, mental fatigue, intellectually slow, difficulty focusing, physical activity). Mean values were calculated for the morning (8 AM), the day (12 AM), the evening (4 PM) and mean per day (mean of 8 AM, 12 AM and 4 PM) were analyzed with score range from 0 to 100. A lower value corresponds to better well-being.
Time Frame: Baseline (week 0), Week 12
Population: ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Hydrocortisone MR Tablet OD - Part A: During the 4-week run-in period prior to the first intervention period during Part A, participants on a twice-a-day (BID) regimen were transferred to a thrice-a-day (TID) regimen while maintaining the same total daily hydrocortisone dose. In the first and second intervention periods during Part A, participants were randomised to novel once daily (OD) treatment with hydrocortisone modified release (MR) tablets 20 to 40 milligram (mg) orally and the treatment continued for 12 weeks and returned every 4 weeks for study drug dispensation.
Arm/Group | Hydrocortisone MR Tablet OD - Part A
Number analyzed (Participants) | 47
scores on a scale | -3.1 (12.1)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A; Test type: Superiority or Other; p = 0.9700, Wilcoxon Signed Rank test

36. Secondary Outcome: Change From Baseline to 6 Months in Diurnal Fatigue Questionnaire for Day Average- Part B
Description: Diurnal fatigue scores (Visual Analog Scale [VAS] scores of energy, relaxed, less alert, moody, mental fatigue, intellectually slow, difficulty focusing, physical activity) were analyzed with score range from 0 to 100. A lower value corresponds to better well-being.
Time Frame: Baseline (week 0), month 6
Population: Part B ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Hydrocortisone MR Tablet OD - Part B (All 6 Months)
Number analyzed (Participants) | 44
scores on a scale | -0.180 (7.943)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part B (All 6 Months); Test type: Superiority or Other; p = 0.2624, Wilcoxon Signed Rank test

37. Secondary Outcome: Comparison on Participant Compliance Between Once Daily and Thrice Daily Therapy - Part A
Description: Compliance was calculated as actual consumption/expected consumption Compliance = (Number of dispensed tablets - Number of returned tablets)/(Number of days during the study period x daily Number of hydrocortisone tablets when taking the ordinary daily dose).
Time Frame: Weeks 4 up to 28
Population: Part A ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: percentage use
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 58 | 58
percentage use | 104.8 (7.5) | 103.1 (13.2)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; Mean difference = 1.28

38. Secondary Outcome: Participant Compliance- Part B
Description: as for outcome 37
Time Frame: Up to Month 6 follow-up
Population: Part B ITT population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: percentage use
Arm/Group | Hydrocortisone MR Tablet OD - Part B (All 6 Months)
Number analyzed (Participants) | 58
percentage use | 102.3 (12.8)

39. Secondary Outcome: Comparison on Participant Preference by Questionnaire Between Once Daily and Thrice Daily Therapy-Part A
Description: Participant Preference Questionnaire consisted of the following set of questions: 1. How large was the benefit with OD compared to TID and the responses were recorded as considerably poorer, somewhat poorer, comparable, large, very large; 2. How strongly concur with the following statement: I prefer novel OD to conventional TID and the responses were recorded as strongly disagree, disagree, neutral, strongly, very strongly; 3. How strongly concur with the following statement: I prefer conventional TID to novel OD and the responses were recorded as strongly disagree, disagree, neutral, strongly, very strongly.
Time Frame: Weeks 16 up to 28
Population: Part A ITT population
Measure: Number; unit: percentage of preference
Groups:
- Hydrocortisone OD Versus TID: Hydrocortisone MR tablets 20 to 40 mg orally OD during Part A of the study. Hydrocortisone tablets 20 to 40 mg orally TID during Part A of the study.
Arm/Group | Hydrocortisone OD Versus TID
Number analyzed (Participants) | 63
percentage of preference
  Benefit compared OD to TID: Considerably poorer | 3.8
  Benefit compared OD to TID: Somewhat poorer | 5.7
  Benefit compared OD to TID: Comparable | 5.7
  Benefit compared OD to TID: Large | 20.8
  Benefit compared OD to TID: Very large | 64.2
  Prefer OD to TID: Strongly disagree | 3.7
  Prefer OD to TID: Disagree | 3.7
  Prefer OD to TID: Neutral | 5.6
  Prefer OD to TID: Strongly | 25.9
  Prefer OD to TID: Very strongly | 61.1
  Prefer TID to OD: Strongly disagree | 39.6
  Prefer TID to OD: Disagree | 35.4
  Prefer TID to OD: Neutral | 12.5
  Prefer TID to OD: Strongly | 4.2
  Prefer TID to OD: Very strongly | 8.3
Statistical Analysis 1: Comparison: Hydrocortisone OD Versus TID; Test type: Superiority or Other; p < 0.0001, Sign test

40. Secondary Outcome: Comparison on 24-hour Urinary Free Cortisol Between Once Daily and Thrice Daily Therapy-Part A
Time Frame: 12 weeks
Population: Part A Safety population consisted of all randomised patients who took at least one dose of study medication. Safety population with participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: nanomoles per 24 hours
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A
Number analyzed (Participants) | 36 | 37
nanomoles per 24 hours | 385.7 (178.8) | 425.9 (278.8)
Statistical Analysis 1: Comparison: Hydrocortisone MR Tablet OD - Part A vs Hydrocortisone Tablet TID - Part A; Test type: Superiority or Other; p = 0.0034, Wilcoxon Signed Rank test; Mean difference = -272.3

ADVERSE EVENTS:
Time Frame: Part A (24 weeks) and Part B (6 months)
Groups:
- Hydrocortisone MR Tablet OD - Part A: Hydrocortisone modified release (MR) tablets 20 to 40 mg orally, once daily (OD) during the 12-week period of Part A.
- Hydrocortisone Tablet TID - Part A: Hydrocortisone tablets 20 to 40 mg orally, thrice daily (TID) during the 12-week period of Part A.
- Hydrocortisone MR Tablet OD - Part B (First 3 Months): Hydrocortisone MR tablets 20 to 40 mg orally, once daily (OD) during the first 3 months of Part B (6 months).
- Hydrocortisone MR Tablet OD - Part B (Second 3 Months): Hydrocortisone MR tablets 20 to 40 mg orally, once daily (OD) during the second 3 months of Part B (6 months).
- Hydrocortisone MR Tablet OD - Part B (All 6 Months): Hydrocortisone MR tablets 20 to 40 mg orally, once daily (OD) during the entire 6-month period of Part B.
Arm/Group | Hydrocortisone MR Tablet OD - Part A | Hydrocortisone Tablet TID - Part A | Hydrocortisone MR Tablet OD - Part B (First 3 Months) | Hydrocortisone MR Tablet OD - Part B (Second 3 Months) | Hydrocortisone MR Tablet OD - Part B (All 6 Months)
Serious Adverse Events (participants affected / at risk) | 6/64 | 2/64 | 2/59 | 4/57 | 6/59
Other Adverse Events (participants affected / at risk) | 29/64 | 25/64 | 12/59 | 16/57 | 23/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocortisone MR Tablet OD - Part A (N=64) | Hydrocortisone Tablet TID - Part A (N=64) | Hydrocortisone MR Tablet OD - Part B (First 3 Months) (N=59) | Hydrocortisone MR Tablet OD - Part B (Second 3 Months) (N=57) | Hydrocortisone MR Tablet OD - Part B (All 6 Months) (N=59)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Surgical and medical procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocortisone MR Tablet OD - Part A (N=64) | Hydrocortisone Tablet TID - Part A (N=64) | Hydrocortisone MR Tablet OD - Part B (First 3 Months) (N=59) | Hydrocortisone MR Tablet OD - Part B (Second 3 Months) (N=57) | Hydrocortisone MR Tablet OD - Part B (All 6 Months) (N=59)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 4 (5)
Fatigue (General disorders) | 8 (10) | 3 (3) | 4 (4) | 2 (2) | 6 (6)
Gastroenteritis (Infections and infestations) | 8 (9) | 2 (2) | 4 (4) | 0 (0) | 4 (4)
Influenza (Infections and infestations) | 8 (8) | 2 (2) | 1 (1) | 4 (4) | 5 (5)
Nasopharyngitis (Infections and infestations) | 7 (9) | 15 (16) | 1 (1) | 6 (6) | 7 (7)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 2 (4) | 5 (7) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicentre publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicentre Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.